CLINICAL TRIAL: NCT05744687
Title: Randomized, Double-blind, Placebo-controlled, Phase II/III Study of SPH4336 Combined With Letrozole vs Placebo Combined With Letrozole in First-line Treatment of HR-positive, HER2-negative Locally Advanced or Metastatic Breast Cancer
Brief Title: Phase II/III Study of SPH4336 Combined With Letrozole vs Placebo Combined With Letrozole in First-line Treatment of Breast Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPH4336-301
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPH4336 Tablets 400mg (Experimental): SPH4336 Tablets； Letrozole tablets
  Interventions: Drug: SPH4336 Tablets 400mg
- SPH4336 Tablets Placebo (Placebo Comparator): SPH4336 Placebo； Letrozole tablets
  Interventions: Drug: SPH4336 Tablets Placebo

INTERVENTIONS:
Drug: SPH4336 Tablets 400mg — SPH4336 Tablets ：Orally, 400mg once a day; 28 days/cycle
  Letrozole tablets ：Orally, 2.5mg once a day; 28 days/cycle
  Arms: SPH4336 Tablets 400mg
Drug: SPH4336 Tablets Placebo — SPH4336 Tablets Placebo：Orally,28 days/cycle
  Letrozole tablets ：Orally, 2.5mg once a day; 28 days/cycle
  Arms: SPH4336 Tablets Placebo

SUMMARY:
This study is designed to evaluate the safety and efficacy of SPH4336 combined with letrozole in first-line treatment of locally advanced or metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily participate in the study, completely understand the study, and voluntarily sign the informed consent form (ICF).
2. Female, ≥ 18 and ≤ 75 years of age at the time of signing the ICF.
3. ECOG（Eastern Cooperative Oncology Group） performance status 0 or 1.
4. Life expectancy ≥ 3 months.
5. Patients with locally advanced or metastatic breast cancer who are unable to receive radical surgeries/other local therapies, with hormone receptor positive and human epidermal growth factor receptor 2 negative confirmed by tumor histopathology and molecular pathology.
6. No previous systemetic therapy for locally advanced or metastatic diseases that cannot receive radical surgeries/other local therapies.
7. At least one measurable lesion as per the Response Evaluation Criteria in Solid Tumors.
8. Postmenopausal or premenopausal/perimenopausal female patients. Premenopausal or perimenopausal women should consent to receive goserelin therapy during the study.
9. Laboratory test results before randomization meet the relevant requirements for organ function.

Exclusion Criteria:

1. Prior treatment with any CDK4/6 （Cyclin dependent kinase）inhibitor.
2. Inflammatory breast cancer.
3. Patients unsuitable for endocrine therapy at the investigator's discretion.
4. History of other malignancies within 5 years prior to the start of study treatment.
5. Patients with known central nervous system metastases.
6. Taking anti-tumor traditional Chinese medicines at the time of signing the ICF.
7. Having undergone a surgery within 28 days prior to the start of study treatment, and hasn't yet recovered from adverse reactions of the surgery.
8. History of myocardial infarction, unstable angina pectoris, severe arrhythmia, and symptomatic congestive heart failure before the start of study treatment; NYHA( New York Heart Association) Class ≥II; QTcF≥ 470 ms; LVEF(Left Ventricular Ejection Fractions)≤ 50%.
9. History of ischemic stroke or severe thromboembolic disease before the start of study treatment.
10. Being receiving potent CYP3A4 inhibitors or inducers at the time of signing the ICF.
11. Hepatitis B surface antigen positive and HBV(Hepatitis B Virus) DNA > 2,000 IU/mL or 104 copies/mL; HCV(hepatitis C virus) antibody positive and HCV RNA positive; or known HIV infection.
12. Patients who participated in a clinical trial and received other investigational drugs within 30 days before the start of study treatment.
13. History of severe anaphylactic diseases, history of severe drug allergy, or known allergy to any ingredient of the investigational product.
14. Presence of diseases or conditions that may impact drug administration or gastrointestinal absorption before the start of study treatment, in the opinion of the investigator, makes them an unsuitable candidate for the study.
15. Uncontrolled infections within 2 weeks before the start of study treatment, in the opinion of the investigator, makes them an unsuitable candidate for the study.
16. Pregnant or lactating women.
17. Known history of substance abuse, excessive drinking, or illegal drug addiction; history of confirmed neurological or mental disorders.
18. Presence of other diseases judged by the investigator that the risks of receiving the study treatment outweigh its benefits, or any other reason for which patients are ineligible for the study as assessed by the investigator and the sponsor.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
response rate (ORR) | Approximately 3years
  tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1.
Progression-free survival (PFS) | Approximately 3years
  from the start date of study treatment to the date of progression disease or death , whichever occurred first.

SECONDARY OUTCOMES:
Cmax | Approximately 3years
  PK (Pharmacokinetics) parameters
Tmax | Approximately 3years
  PK (Pharmacokinetics) parameters
Disease control rate (DCR) | Approximately 3years
  DCR was defined as the percentage of patients who have achieved complete response, partial response and stable disease.
Duration of remission (DOR) | Approximately 3years
  DOR was defined for participants who had an objective response as the time from the first occurrence of a documented unconfirmed response to the date of disease progression per RECIST v1.1 or death from any cause.
Overall Survival (OS) | Approximately 8years
  Determination of the overall survival times of all patients.
Incidence of Adverse event | Approximately 3years
  Safety and tolerability

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Affiliated Cancer Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - AnYang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The Second Norman Bethune Hospital of Jilin Univer, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Peking University Cancer Hospital, Beijing